CLINICAL TRIAL: NCT05478837
Title: PNOC018 A Phase 1 Clinical Trial of Autologous T Cells Expressing a TCR Specific for H3.3K27M With Inhibition of Endogenous TCR (KIND T Cells) in HLA-A*0201-positive Participants With H3.3K27M-positive Diffuse Midline Gliomas
Brief Title: Genetically Modified Cells (KIND T Cells) for the Treatment of HLA-A*0201-Positive Patients With H3.3K27M-Mutated Glioma
Acronym: PNOC018
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The V Foundation (Other); Parker Institute for Cancer Immunotherapy (Other); Alliance for Cancer Gene Therapy (Other)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210813; NCI-2022-05420 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); PICI0029 (Other: Parker Institute for Cancer Immunotherapy)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: Autologous T Cells; KIND T Cells; HLA-A*0201-Positive
MeSH Terms: interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (KIND T cells, cyclophosphamide, fludarabine) (Experimental): Patients receive fludarabine IV on days -4, -3, and -2 and cyclophosphamide IV on day -2 in the absence of disease progression or unacceptable toxicity for the conditioning regimen. Patients also receive KIND T cells IV at dose level 1 (2 x 106 dextramer®+ CD8+ cells/kg) on day 0. If no DLTs are reported, newly enrolling participants may receive dose level 2 of KIND T cells on day 0.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Autologous Anti-H3.3K27M TCR-expressing T-cells

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan; Cycloblastin
Drug: Fludarabine — Given IV
  Other Names: Fludara
Biological: Autologous Anti-H3.3K27M TCR-expressing T-cells — Given IV
  Other Names: KIND T cells

SUMMARY:
This phase I, first-in-human trial tests the safety, side effects, and best dose of genetically modified cells called KIND T cells after lymphodepletion (a short dose of chemotherapy) in treating patients who are HLA-A*0201-positive and have H3.3K27M-mutated diffuse midline glioma. KIND T cells are a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory into KIND T cells so they will recognize certain markers found in tumor cells. Drugs such as cyclophosphamide and fludarabine are chemotherapy drugs used to decrease the number of T cells in the body to make room for KIND T cells. Giving KIND T cells after cyclophosphamide and fludarabine may be more useful against cancer compared to the usual treatment for patients with H3.3K27M-mutated diffuse midline glioma (DMG).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of a single intravenous (IV) infusion of autologous anti-H3.3K27M T-cell receptor (TCR) -expressing T-cells (KIND T cells) in HLA-A*0201+ participants with H3.3K27M+ diffuse midline gliomas.

II. To determine the feasibility of a single intravenous (IV) infusion of KIND T cells in HLA-A*0201+ participants with H3.3K27M+ diffuse midline gliomas.

SECONDARY OBJECTIVES:

I. To evaluate manufacturing feasibility of KIND T cells. II. To characterize KIND T cells with respect to their expansion and persistence.

EXPLORATORY OBJECTIVES:

I. To describe antitumor responses and survival after infusion of KIND T cells

II. To explore the association of tumor and immune biomarkers including but not limited to characterization of KIND T cells in blood and tumor samples with clinical endpoints and/or AEs

III. To assess Health-Related Quality of Life (HRQoL) in patients newly diagnosed with HLA-A*0201+ H3.3K27M+ DMG.

IV. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures in the context of race ethnicity and other health related social risks.

V. To assess on therapy toxicity in the context of race, ethnicity and other health related social risks.

OUTLINE: This is a dose-escalation study of KIND T cells.

CONDITIONING REGIMEN: Patients receive fludarabine intravenously (IV) on days -4, -3, and -2 and cyclophosphamide IV on day -2 in the absence of disease progression or unacceptable toxicity.

T CELL THERAPY: Patients receive KIND T cells IV over 10 minutes on day 0.

After completion of study treatment, patients are followed up at day 1, 3, 7, 10, 14, 21, and 28, weeks 8-24 and 28-92, months 24-36, and then yearly until year 15.

ELIGIBILITY:
Inclusion Criteria:

* Participants 2 to 25 years of age inclusive, at the time of signing the informed consent. The first two participants will be 12-25 years of age.
* Male participants of impregnate potential must agree to use contraception, during the study and for at least 6 months after the last study intervention and refrain from donating sperm during this period.
* Female participants of childbearing potential must agree to follow the contraceptive guidance, during the study and for at least 6 months after the last study intervention.
* Females of childbearing potential must have a negative serum or urine pregnancy test within 14 days of receiving study interventions.
* CNS reservoir such as Ommaya catheter must be in place.
* Patients must be enrolled on PNOC COMP prior to enrollment on PNOC018 if PNOC COMP is open to accrual at the enrolling institution.
* Participants with DMG who are positive for the H3.3K27M mutation (positive testing from a Clinical Laboratory Improvement Amendments (CLIA) laboratory required or equivalent) and who completed at least standard radiation therapy.
* All participants must test positive for HLA-A*0201 (positive testing from a CLIA or equivalent laboratory required). Other HLA-A2 subtypes are excluded.
* All participants must consent for tumor tissue (fresh or archival) for biomarker analysis if available.
* All participants must have evaluable or measurable disease at the time of consent.
* All participants must be either off systemic steroids or be on a stable or declining dose of dexamethasone (maximum dose of 0.1 mg/kg/day or 4 mg/day) at the time of enrollment.
* Participants must not have received any bone marrow transplants for the treatment of their tumor.
* Participants must discontinue all anti-cancer agents and radiotherapy and, must have recovered from significant acute toxic effects of prior therapies.

  * Chemotherapy/biologic therapy: All cytotoxic chemotherapy/biologic therapy must be discontinued ≥ 7 days prior to enrollment.
  * Immunotherapy: The last dose of anti-tumor antibody therapy must be at least 3 half-lives or 30 days, whichever is shorter, from the time of enrollment.
* All participants must have adequate organ function.
* Adequate bone marrow function is defined as:

  * Peripheral absolute neutrophil account 1000/mm^3 and
  * Platelet count 100,000/mm^3 (transfusion dependent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Absolute lymphocyte count >= 500/µL or CD3 count of >= 150/µL
* Adequate renal function is defined as:
* Creatinine clearance or radioisotope glomerular filtration rate >= 70 mL/min/1.73 m^2 or
* Maximum serum creatinine based on age/gender as follows:

  * 3 to < 6 years =< 0.8 mg/dL (male and female)
  * 6 to < 10 years =< 1.0 mg/dL (male and female)
  * 10 to < 13 years =< 1.2 mg/dL (male and female)
  * 13 to < 16 years =< 1.5 mg/dL (male) and 1.4 mg/dL (female)
  * >= 16 years =< 1.7 mg/dL (male) and 1.4 mg/dL (female)
* Adequate liver function is defined as:

  * Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age and
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN and
  * Serum albumin >= 2 g/dL
* Participants with a history of congestive heart failure at risk because of underlying cardiovascular disease or exposure to cardiotoxic drugs must have adequate cardiac function as clinically indicated. Only order ECHO and EKG for patients with history of cardiac toxicity.

  * (QTc) =< 480 ms
  * Injection fraction >= 45% by echocardiogram
* Adequate pulmonary function is defined as no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and pulse oximetry > 92% while breathing room air
* Adequate neurologic function is defined as a well-controlled seizure disorder and performance status (Lansky < 16 years and Karnofsky >= 16 years) that is at least 60.
* Informed consent: Capable of giving signed informed consent or assent depending on participant age as appropriate which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Assent will be obtained when appropriate based on the subjects age.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Participants with MRI or clinical evidence of uncontrolled tumor mass effect; the assessment of mass effect should be made by the study investigators prior to any planned KIND T cell treatment. Pre-infusions MRI will need to be reviewed by the study investigators prior to dosing. Participants with an assessment score >= 3 will be excluded, based on Table 4 in section 3.8.2
* Participants with a known disorder that affects their immune system such as HIV or hepatitis B or C, or an autoimmune disorder requiring systemic cytotoxic or immunosuppressive therapy. Participants who are currently using inhaled, intranasal, ocular, topical, or other non-oral or non-IV steroids are not necessarily excluded from the study.
* Participants who have received prior solid organ or bone marrow transplantation.
* Participants with uncontrolled infection.
* Female participants of childbearing potential must not be pregnant or breast-feeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Untreated symptomatic hydrocephalus determined by treating physician.
* Participants who are unable to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.
* Participants who are currently receiving another investigational drug.
* Participants who are co-enrolled on another investigational protocol.
* Participants who are currently receiving other anticancer agents (bevacizumab used to treat tumor mass effect will not constitute an exclusion; at time of enrollment participants need to be off bevacizumab and will need to be discussed with the study team).

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Up to 28 days following infusion of autologous anti-H3.3K27M TCR-expressing T-cells (KIND T cells)
  To determine the safety and tolerability of a single intravenous (IV) infusion of KIND T cells in HLA A*0201+ participants with H3.3K27M+ diffuse midline gliomas
Percent of successfully manufactured KIND T cells | Up to 24 months
  To determine feasibility of a single intravenous (IV) infusion of KIND T cells in HLA A*0201+ participants with H3.3K27M+ diffuse midline gliomas

SECONDARY OUTCOMES:
Percentage of participants who receive KIND T cells | Up to 12 months
  The percentage of participants who received KIND T cell infusions will be reported. If the manufacturing of T-cell product is not successful because it does not meet release criteria, the participant will have the choice of a second apheresis for a second manufacturing process
Duration of KIND T cells in-vivo persistence | Up to 12 months
  The duration of KIND T cells in-vivo persistence will be estimated using Kaplan-Meier techniques. In addition, the persistence of KIND T cells will be evaluated for each participant for up to 12 months or until any 2 sequential negative tests documenting loss of KIND T cells in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Principal Investigator — University of California, San Francisco; Hideho Okada, MD, PhD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification.
Supporting Information: Study Protocol